CLINICAL TRIAL: NCT03266211
Title: Antitetanus Vaccination for People Older Than 65 Years in the Auvergne-Rhône-Alpes (France) Region Depending on the Demographic and Medical Practice of Their Medical Practitioner.
Brief Title: Antitetanus Vaccination for People Older Than 65 Years.
Acronym: VAT65
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0375
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2017-08

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: People older than 65 years in the Auvergne-Rhônes-Alpes region who are consulting their general practitioner.
  Interventions: Other: Questionnaire Patients
- General practitioner: General practitioner of the Auvergne-Rhônes-Alpes region
  Interventions: Other: Questionnaire General practitioner

INTERVENTIONS:
Other: Questionnaire Patients — Patient will have to answer a quiz which is about their vaccination against tetanus.
  Groups: Patients
Other: Questionnaire General practitioner — General practitioner will have to answer a quiz which is about their medical practice concerning vaccination against tetanus.
  Groups: General practitioner

SUMMARY:
In the last ten years, more than one hundred generalized tetanus cases were declared in France. Most of them were affecting people older than 70 years with an important mortality (around 28%). It is know that the only way to protect ourselves from this disease is the vaccination. In France tetanus vaccination is mandatory since 1940.

Nowaday none study looked specifically for the vaccination of people older than 65 years. The hypothesis is: there is a difference in the tetanus vaccination coverage for people older than 65 years depending on the demographic and medical practice of their general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years consulting their attending physician in and who agreed to participate in the study.
* The doctors included are general practitioners located in a liberal office in the "Auvergne Rhône Alpes" region for which the URPS ("Union régional des Professionnels de Santé") has an email address.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be all patients older than 65 years who are consulting their general practitioner and accepting to participate to the study. And their general practitioner.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Tetanus vaccination coverage | About 5 minutes
  Patient will have to answer a quiz which is about their vaccination against tetanus.

CONTACTS AND LOCATIONS:
Locations (1):
- Service Urgence et Réanimation Pédiatrique Hôpital Femme Mère Enfant Groupement Hospitalier Est, Bron, France

IPD SHARING:
Plan to Share IPD: No